CLINICAL TRIAL: NCT03945539
Title: An Open-label, Fixed-sequence, Drug-drug Interaction Study to Evaluate the Effect of Itraconazole on the Pharmacokinetics of JNJ-56136379 in Healthy Adult Participants
Brief Title: A Study to Evaluate the Effect of Itraconazole on JNJ-56136379 in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Sciences Ireland UC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108614; 2019-000966-39 (EudraCT Number); 56136379HPB1008 (Other: Janssen Sciences Ireland UC)
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — JNJ-56136379; Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JNJ-56136379 and Itraconazole (Experimental): Participants will receive a single dose of JNJ-56136379 on Day 1 in Treatment Period 1 and itraconazole 200 mg once daily for 21 days starting on Day 34 along with a single dose of JNJ 56136379 on Day 38 in Treatment Period 2. JNJ-56136379 intake in Treatment Period 1 and the first intake of itraconazole in Treatment Period 2 will be separated by a washout period of at least 33 days. Study drug (JNJ-56136379 and itraconazole) intakes will be taken orally and under fed conditions.
  Interventions: Drug: JNJ-56136379; Drug: Itraconazole

INTERVENTIONS:
Drug: JNJ-56136379 — Participants will receive JNJ-56136379 orally on Day 1 in Treatment Period 1 and on Day 38 in Treatment Period 2.
Drug: Itraconazole — Participants will receive 200 mg of itraconazole once daily orally for 21 days starting on Day 34.

SUMMARY:
The main purpose of this study is to assess the effect of itraconazole at steady-state on a single-dose pharmacokinetic (PK) of JNJ-56136379 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy on the basis of physical examination, clinical laboratory tests, medical history, and vital signs performed at screening. If there are abnormalities, the participant may be included only if the investigator judges the abnormalities to be not clinically significant or to be appropriate and reasonable for the population under study. This determination must be recorded in the participant's source documents and initialed by the investigator
* Must not use nicotine-containing substances including tobacco products for at least 3 months prior to screening and during the study
* A woman of childbearing potential must have a negative highly sensitive serum pregnancy test (beta-human chorionic gonadotropin) at screening and a negative urine pregnancy test at Day -1 of the first treatment period
* Body mass index (weight kilogram [kg]/height^2 meter [m]^2) between 18.0 and 30.0 kg/m^2 (inclusive), and body weight not less than 50.0 kg
* Blood pressure (after the participant is supine for 5 minutes) between 90 and 140 millimeters of Mercury (mmHg) systolic, inclusive, and no higher than 90 mmHg diastolic. If blood pressure is out of range, up to 2 repeated assessments are permitted

Exclusion Criteria:

* History of cardiac arrhythmias (example [e.g.], tachycardia at rest), history of risk factors for Torsade de Pointes syndrome (e.g., hypokalemia, family history of long QT Syndrome) at screening
* Any evidence of heart block or bundle branch block at screening
* Any current, or history of, clinically significant skin disease at screening requiring intermittent or chronic treatment (at the investigator's discretion) such as, but not limited to, dermatitis, eczema, drug rash, psoriasis, food allergy, and urticaria
* Known allergies, hypersensitivity, or intolerance to JNJ-56136379 or itraconazole or its excipients at screening
* History of clinically significant drug allergy at screening such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous studies with experimental drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2019-10-04 (Actual); Study Completion 2019-10-04 (Actual)

PRIMARY OUTCOMES:
Period 1: Area Under the Plasma Analyte Concentration Versus Time Curve From time 0 to 72 hours Postdose (AUC [0-72 hours]) of JNJ-56136379 | Predose (Day 1), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours postdose on Day 4
  AUC [0-72 hours] is defined as area under the plasma analyte concentration versus time curve from time 0 to 72 hours postdose.
Period 2: Area Under the Plasma Analyte Concentration Versus Time Curve From time 0 to 72 hours Postdose (AUC [0-72 hours]) of JNJ-56136379 | Predose (Day 38), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours postdose on Day 41
  AUC [0-72 hours] is defined as area under the plasma analyte concentration versus time curve from time 0 to 72 hours postdose.
Period 1: Area Under the Plasma Analyte Concentration Versus Time Curve From Time 0 to 408 Hours Posdose AUC [0-408 hours] of JNJ-56136379 | Predose (Day 1), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 and 408 hours postdose on Day 18
  AUC [0-408 hours] is defined as area under the plasma analyte concentration versus time curve from time 0 to 408 hours postdose.
Period 2: Area Under the Plasma Analyte Concentration Versus Time Curve From Time 0 to 408 Hours Posdose AUC [0-408 hours] of JNJ-56136379 | Predose (Day 38), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 144, 168, 216, 336 and 408 hours postdose on Day 55
  AUC [0-408 hours] is defined as area under the plasma analyte concentration versus time curve from time 0 to 408 hours postdose.
Period 1: Maximum Observed Plasma Analyte Concentration of JNJ-56136379 | Predose (Day 1), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336 and 408 hours postdose on Day 18
  Cmax is defined as maximum observed plasma analyte concentration.
Period 2: Maximum Observed Plasma Analyte Concentration of JNJ-56136379 | Predose (Day 38), 0, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72, 120, 144, 168, 216, 336 and 408 hours postdose on Day 55
  Cmax is defined as maximum observed plasma analyte concentration.

SECONDARY OUTCOMES:
Number of Participants with Adverse Event as Measure of Safety and Tolerability | Approximately 100 Days
  An Adverse Event is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Sciences Ireland UC Clinical Trial, Study Director — Janssen Sciences Ireland UC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency